CLINICAL TRIAL: NCT05193058
Title: Description of Lung Transplant Patients With Microbiologically Documented Stenotrophomonas Maltophilia Pneumonia and Impact of Treatment on Outcome
Acronym: STENO_SOT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: STENO_SOT
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Transplantation Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Stenotrophomonas maltophilia is a multi-resistant Gram-negative bacillus and is an opportunistic pathogen. Stenotrophomonas maltophilia infections are associated with a significant morbidity and mortality, particularly in immunocompromised patients. The mortality of infections (bacteremia, pneumonia) related to Stenotrophomonas maltophilia is variable and is estimated between 21 and 69%. Stenotrophomonas maltophilia pneumopathies have been mainly described in patients hospitalized in intensive care and benefiting from mechanical ventilation. The existence of immunosuppression seems to be a risk factor for the transition from Stenotrophomonas maltophilia pulmonary colonization to Stenotrophomonas maltophilia pulmonary infection. The reference treatment for Stenotrophomonas maltophilia-associated pneumonia is the combination of trimethoprim and sulfamthoxazole, a molecule that lung transplant patients routinely receive as a preventive treatment for Pneumocysitis jirovecii infection. There is no consensus on the value of routine dual-antibiotic therapy, and it varies from one center to another and from one country to another.

The main objective is to compare the clinical-microbiological evolution of lung transplant patients treated for Stenotrophomonas maltophilia pneumopathy according to the prescription of a mono- or bi-antibiotherapy.

The secondary objective is to evaluate the resistance rate of Stenotrophomonas maltophilia strains isolated from respiratory samples according to the anti-pneumocystis prophylactic molecule received by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patient whose age ≥ 18 years
* Patient who has received a lung (mono or bi-pulmonary) or heart-lung transplant
* Patient with documented pneumopathy (clinico-radiological definition) (positive respiratory specimen for Stenotrophomonas maltophilia)
* French speaking patient

Exclusion Criteria:

* Patient under guardianship or curatorship
* Patient deprived of liberty
* Patient under court protection
* Patient objecting to the use of his data for this research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients managed for Stenotrophomonas maltophilia pneumonia following a lung or heart-lung transplant between 01/01/2011 and 01/01/2021
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-11-22 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical-microbiological course of lung transplant patients treated for Stenotrophomonas maltophilia pneumonia | Day 1
  This outcome corresponds to the comparison of mortality and recurrence rates of Stenotrophomonas maltophilia pneumonia according to the prescription of mono- or dual-antibiotic therapy.

SECONDARY OUTCOMES:
Resistance rate of Stenotrophomonas maltophilia strains | Day 1
  This outcome corresponds to the Trimethorpime/sulfamethoxazole resistance rate of Stenotrophomonas maltophilia strains.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit PILMIS, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Denton M, Kerr KG. Microbiological and clinical aspects of infection associated with Stenotrophomonas maltophilia. Clin Microbiol Rev. 1998 Jan;11(1):57-80. doi: 10.1128/CMR.11.1.57. PMID 9457429
- [Background] Senol E, DesJardin J, Stark PC, Barefoot L, Snydman DR. Attributable mortality of Stenotrophomonas maltophilia bacteremia. Clin Infect Dis. 2002 Jun 15;34(12):1653-6. doi: 10.1086/340707. Epub 2002 May 24. PMID 12032905
- [Background] Prates M, Fernandes F, Proenca F, Mussa Y, Tavares A, Pereira A. Oral Infection Caused by Stenotrophomonas maltophilia: A Rare Presentation of an Emerging Opportunistic Pathogen. Case Rep Infect Dis. 2020 Jan 29;2020:6346120. doi: 10.1155/2020/6346120. eCollection 2020. PMID 32082659
- [Background] Hashimoto T, Komiya K, Fujita N, Usagawa Y, Yamasue M, Umeki K, Ando M, Nureki SI, Hiramatsu K, Kadota JI. Risk factors for 30-day mortality among patients with Stenotrophomonas maltophilia bacteraemia. Infect Dis (Lond). 2020 Jun;52(6):440-442. doi: 10.1080/23744235.2020.1734653. Epub 2020 Mar 3. No abstract available. PMID 32122208
- [Background] Saugel B, Eschermann K, Hoffmann R, Hapfelmeier A, Schultheiss C, Phillip V, Eyer F, Laugwitz KL, Schmid RM, Huber W. Stenotrophomonas maltophilia in the respiratory tract of medical intensive care unit patients. Eur J Clin Microbiol Infect Dis. 2012 Jul;31(7):1419-28. doi: 10.1007/s10096-011-1459-8. Epub 2011 Nov 7. PMID 22057419
- [Background] Flamm RK, Shortridge D, Castanheira M, Sader HS, Pfaller MA. In Vitro Activity of Minocycline against U.S. Isolates of Acinetobacter baumannii-Acinetobacter calcoaceticus Species Complex, Stenotrophomonas maltophilia, and Burkholderia cepacia Complex: Results from the SENTRY Antimicrobial Surveillance Program, 2014 to 2018. Antimicrob Agents Chemother. 2019 Oct 22;63(11):e01154-19. doi: 10.1128/AAC.01154-19. Print 2019 Nov. PMID 31427295
- [Background] Chang YT, Lin CY, Chen YH, Hsueh PR. Update on infections caused by Stenotrophomonas maltophilia with particular attention to resistance mechanisms and therapeutic options. Front Microbiol. 2015 Sep 2;6:893. doi: 10.3389/fmicb.2015.00893. eCollection 2015. PMID 26388847